CLINICAL TRIAL: NCT01143116
Title: Reduction of Bacteriuria in Subjects Practicing Intermittent Catheterization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wellspect HealthCare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: YA-ABC-0003
Record Dates: First submitted 2010-06-09; First posted 2010-06-14 (Estimated); Results first posted 2022-05-03 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-05

CONDITIONS: Bacteriuria
MeSH Terms: conditions — Bacteriuria

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Study subjects, study personnel and laboratory conducting the cultivations and analyses were blinded to the investigational products. The products had the same packaging and visual appearance. The treatment code was never broken during the study.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Catheter A (Experimental): Catheterization with Catheter A, which releases silver ions into the urethra and urinary bladder upon catheterization,.
  After activation in the wetting solution the coating retains water creating a smooth liquid surface around the catheter.The products are intended for single use. No additional lubricant were used.
  The subject will be treated with investigational products during 24 hours. During this period the subject will be catheterized with the study catheter at six occasions (every 4 hours).
  Interventions: Device: Silver-nitrate coated catheter ("Catheter A")
- Catheter B (Experimental): Catheterization with Catheter B, which releases both silver ions and degradable silver particles.. After activation in the wetting solution the coating retains water creating a smooth liquid surface around the catheter.The products are intended for single use. No additional lubricant were used.
  The subject will be treated with investigational products during 24 hours. During this period the subject will be catheterized with the study catheter at six occasions (every 4 hours).
  Interventions: Device: Degradable silver particle-coated catheter ("Catheter B")

INTERVENTIONS:
Device: Silver-nitrate coated catheter ("Catheter A") — Catheter A releases silver ions into the urethra and urinary bladder upon catheterization.
  Arms: Catheter A
Device: Degradable silver particle-coated catheter ("Catheter B") — Catheter B releases both silver ions and degradable silver particles into the urethra and urinary bladder upon catheterization.
  Arms: Catheter B

SUMMARY:
The main objective is to investigate two types of antibacterial catheters regarding their antibacterial efficacy. The study will investigate if silver added to the coating of a urinary catheter exerts antibacterial activity that will have an impact on bacteria quantity in the urine bladder among users of intermittent catheterization.

DETAILED DESCRIPTION:
The study was designed as a prospective, randomized, double-blind, single-site study of 24 hours use of a silver coated antibacterial catheter, and 24 hours follow up, in subjects practicing intermittent catheterization.

Twenty male and female subjects using intermittent catheterization, having a confirmed significant bacteriuria were included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent
* Female/male aged 18 years and over
* Practicing intermittent catheterization at least 4 times daily for at least 6 weeks
* A minimum of 104 CFU of bacteriuria

Exclusion Criteria:

* Ongoing, symptomatic UTI at enrollment
* Known urethral stricture
* Basic tumorous disease
* Previous prostate surgery
* Subjects known to be immunocompromised e.g. HIV or diabetes
* Treatment with antibiotics and/or intravesical antiseptics for the past 30 days before study start
* Involvement in the planning and conduct of the study (applies to both Astra Tech staff or staff at the study site)
* Pregnancy or breast feeding
* Previous enrolment or randomisation of treatment in the present study
* Participation in a clinical study that possibly might interfere with the present study, as deemed by the investigator
* Severe non-compliance to protocol as judged by the investigator and/or Astra Tech

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-11; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Waigh El Masri, Mr, Principal Investigator — The Robert Jones and Agnes Hunt Orthopaedic and District Hospital NHS Trust
Locations (1):
- The Robert Jones and Agnes Hunt Orthopaedic and District Hospital NHS Trust, Oswestry, Shropshire, United Kingdom

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Catheter A | Catheter B
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Catheter A | Catheter B | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (8) | 40 (8) | 44 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 9 | 8 | 17
Region of Enrollment [Number; unit: participants]
  Sweden | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Total Bacteria Count Change From Baseline and After 24 Hours.
Description: Change from baseline (urine sample immediately before first catheterization with study product) and after 24 hours of intermittent catheterization with the randomised study catheter.
Time Frame: Baseline and after 24 hours
Population: ITT
Measure: Mean (Standard Deviation); unit: CFU/mL
Arm/Group | Catheter A | Catheter B
Number analyzed (Participants) | 10 | 10
CFU/mL | -62519 (9710767) | 57448 (9810360)
Statistical Analysis 1: Comparison: Catheter A; Test type: Other; p = 0.6250, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Catheter B; Test type: Other; p = 0.7500, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Total Bacteria Count Change From Baseline and After 48 Hours.
Description: Change from baseline (urine sample immediately before first catheterization with study product) and after 48 hours of intermittent catheterization.
  After the baseline sample the subject had 24 hours with study randomized catheter and then changed to 24 hours on non-study sterile intermittent catheterization.
Time Frame: Baseline and after 48 hours
Population: ITT
Measure: Mean (Standard Deviation); unit: CFU/mL
Arm/Group | Catheter A | Catheter B
Number analyzed (Participants) | 10 | 10
CFU/mL | -1980704 (6599515) | 2072657 (11673736)
Statistical Analysis 1: Comparison: Catheter A; Test type: Other; p = 0.8750, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Catheter B; Test type: Other; p = 0.6250, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Total Bacteria Count Change From Baseline and After 7-14 Days.
Description: Change from baseline and after 7-14 days. Change from baseline (urine sample immediately before first catheterization with study product) to after 7-14 days.
Time Frame: Baseline and after 7-14 days
Population: ITT
Measure: Mean (Standard Deviation); unit: CFU/mL
Arm/Group | Catheter A | Catheter B
Number analyzed (Participants) | 10 | 10
CFU/mL | 12477797 (10769480) | 18650000 (6851389)
Statistical Analysis 1: Comparison: Catheter A; Test type: Other; p = 0.0254, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Catheter B; Test type: Other; p = 0.0039, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Escherichia Coli Mean Bacteria Count Change From Baseline to 12 Hours
Description: Escherichia coli mean bacteria count change from baseline (subjects with positive values) to after 12 hours.
  Baseline (urine sample immediately before first catheterization with study product) and then at 12 hours of study catheter use.
Time Frame: After first catheterization with study product and after 12 hours
Population: Subjects with positive values
Measure: Mean (Standard Deviation); unit: CFU/mL
Arm/Group | Catheter A | Catheter B
Number analyzed (Participants) | 4 | 5
CFU/mL | 0 (0) | 74500 (166587)
Statistical Analysis 1: Comparison: Catheter A; Test type: Other; p = 1.0, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Catheter B; Test type: Other; p = 1.0000, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Escherichia Coli Mean Bacteria Count Change From Baseline to 24 Hours
Description: Escherichia coli mean bacteria count change from baseline (subjects with positive values).
  Baseline (urine sample immediately before first catheterization with study product) and then at 24 hours of study catheter use.
Time Frame: After first catheterization with study product and after 24 hours
Population: Subjects with positive values
Measure: Mean (Standard Deviation); unit: CFU/mL
Arm/Group | Catheter A | Catheter B
Number analyzed (Participants) | 4 | 5
CFU/mL | 5113750 (10227500) | -4124000 (9221544)
Statistical Analysis 1: Comparison: Catheter A; Test type: Other; p = 1.0, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Catheter B; Test type: Other; p = 1.0000, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Enterococcus Faecalis Mean Bacteria Count Change From Baseline to 12 Hours
Description: Enterococcus faecalis mean bacteria count change from baseline (subjects with positive values).
  Baseline (urine sample immediately before first catheterization with study product) and then at 12 hours of study catheter use.
Time Frame: After first catheterization with study product and after 12 hours
Population: Subjects with positive values
Measure: Mean (Standard Deviation); unit: CFU/mL
Arm/Group | Catheter A | Catheter B
Number analyzed (Participants) | 2 | 1
CFU/mL | 333 (612) | 20997300
Statistical Analysis 1: Comparison: Catheter A; Test type: Other; p = 1.0000, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Enterococcus Faecalis Mean Bacteria Count Change From Baseline to 24 Hours
Description: Enterococcus faecalis mean bacteria count change from baseline (subjects with positive values).
  Baseline (urine sample immediately before first catheterization with study product) and then at 24 hours of study catheter use.
Time Frame: After first catheterization with study product and after 24 hours
Population: Subjects with positive values
Measure: Mean (Standard Deviation); unit: CFU/mL
Arm/Group | Catheter A | Catheter B
Number analyzed (Participants) | 2 | 1
CFU/mL | -51498 (73684) | 20999983
Statistical Analysis 1: Comparison: Catheter A; Test type: Other; p = 1.0000, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Urine Silver Concentration Change From Baseline to 24 Hours
Description: Urine silver concentration change from baseline excluding five subjects with extreme outlier values at baseline due to laboratory error during analysis and all subjects presented normal values during study follow up.
  Samples for analysis of silver concentration in urine were collected at baseline, after last catheterization with investigational product (at the very end of day 2) at the last catheterization at day 3 and at study termination (at 7-14 days).
Time Frame: Baseline to 24 hours
Population: Per protocol, excluding five subjects with extreme outlier values at baseline due to laboratory error during analysis and all subjects presented normal values during study follow up.
Measure: Mean (Standard Deviation); unit: nmol Ag/mmol creatinine
Arm/Group | Catheter A | Catheter B
Number analyzed (Participants) | 7 | 8
nmol Ag/mmol creatinine | 5.15 (9.70) | 6.20 (5.26)
Statistical Analysis 1: Comparison: Catheter A; Test type: Other; p = 0.0313, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Catheter B; Test type: Other; p = 0.0078, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Urine Silver Concentration Change From Baseline and After 48 Hours
Description: as for outcome 8
Time Frame: After first catheterization with study product and after 48 hours
Population: Per protocol excluding five subjects with extreme outlier values at baseline due to laboratory error during analysis and all subjects presented normal values during study follow up.
Measure: Mean (Standard Deviation); unit: nmol Ag/mmol creatinine
Arm/Group | Catheter A | Catheter B
Number analyzed (Participants) | 7 | 8
nmol Ag/mmol creatinine | -0.02 (0.11) | -0.02 (0.12)
Statistical Analysis 1: Comparison: Catheter A; Test type: Other; p = 0.7188, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Catheter B; Test type: Other; p = 0.6406, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Urine Silver Concentration Change From Baseline to 7-14 Days
Description: as for outcome 8
Time Frame: At baseline and after 7-14 days
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: nmol Ag/mmol creatinine
Arm/Group | Catheter A | Catheter B
Number analyzed (Participants) | 7 | 8
nmol Ag/mmol creatinine | 0.39 (0.53) | 0.10 (0.24)
Statistical Analysis 1: Comparison: Catheter A; Test type: Other; p = 0.4375, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Catheter B; Test type: Other; p = 0.2969, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Blood Silver Concentration Change From Baseline and After 24 Hours
Description: Samples for analysis of silver concentration in blood were collected at baseline, after last catheterization with investigational product (at the very end of day 2) at the last catheterization at day 3 and at study termination (at 7-14 days).
Time Frame: After first catheterization with study product and after 24 hours
Population: ITT
Measure: Mean (Standard Deviation); unit: nmol Ag/L
Arm/Group | Catheter A | Catheter B
Number analyzed (Participants) | 10 | 10
nmol Ag/L | -.02 (0.28) | 0.39 (0.22)
Statistical Analysis 1: Comparison: Catheter A; Test type: Other; p = 0.5391, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Catheter B; Test type: Other; p = 0.0010, Wilcoxon (Mann-Whitney)

12. Secondary Outcome: Blood Silver Concentration Change From Baseline and After 48 Hours
Description: as for outcome 11
Time Frame: After first catheterization with study product and after 48 hours
Population: ITT
Measure: Mean (Standard Deviation); unit: nmol Ag/L
Arm/Group | Catheter A | Catheter B
Number analyzed (Participants) | 10 | 10
nmol Ag/L | 0.02 (0.48) | 0.27 (0.25)
Statistical Analysis 1: Comparison: Catheter A; Test type: Other; p = 0.4766, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Catheter B; Test type: Other; p = 0.0068, Wilcoxon (Mann-Whitney)

13. Secondary Outcome: Blood Silver Concentration Change From Baseline and After 7-14 Days
Description: as for outcome 11
Time Frame: After first catheterization with study product and after 7-14 days
Population: ITT
Measure: Mean (Standard Deviation); unit: nmol Ag/L
Arm/Group | Catheter A | Catheter B
Number analyzed (Participants) | 10 | 10
nmol Ag/L | 0.31 (0.54) | -0.04 (0.61)
Statistical Analysis 1: Comparison: Catheter A; Test type: Other; p = 0.0625, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Catheter B; Test type: Other; p = 0.4180, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 3 days. The study was performed during 3 days starting with a wash out during one day, then the randomized study product was used for one day, ending with a wash out day with a non-study product.
Description: Adverse events/adverse device effects were collected during all three days but only observed and reported during the 24 hours use of the test catheters. No adverse events/adverse device effects were observed during the time (24 h) prior to use of the test catheters or after (24h).
  Observed by the Study personnel or spontaneously reported from the subject.
Arm/Group | Catheter A | Catheter B
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 3/10 | 3/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Catheter A (N=10) | Catheter B (N=10)
Fever (General disorders) | 0 (0) | 1 (1)
Headache (General disorders) | 0 (0) | 2 (2)
Rash in the right leg (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Frequency of micturation increased (Renal and urinary disorders) | 1 (1) | 0 (0)
Wrist pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Symptoms of urinary tract infection (Renal and urinary disorders) | 1 (1) | 0 (0)
Sensation of preassure in the bladder (Renal and urinary disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No